CLINICAL TRIAL: NCT03736967
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study to Assess the Efficacy and Safety of REGN3500 Monotherapy and Combination of REGN3500 Plus Dupilumab in Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Efficacy and Safety of REGN3500 Monotherapy and Combination of REGN3500 Plus Dupilumab in Adult Patients With Moderate-to-Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3500-AD-1798; 2018-001543-30 (EudraCT Number)
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: Moderate; Severe
MeSH Terms: conditions — Dermatitis, Atopic; Lymphoma, Follicular | interventions — itepekimab; dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- REGN3500 (Experimental)
  Interventions: Drug: REGN3500
- Dupilumab (Experimental)
  Interventions: Drug: Dupilumab
- Combo (Experimental)
  Interventions: Drug: REGN3500 + Dupilumab Combo
- Placebo (Experimental)
  Interventions: Drug: REGN3500; Drug: Dupilumab; Drug: Placebo

INTERVENTIONS:
Drug: REGN3500 — Administered subcutaneous (SC) every 2 weeks (q2w)
  Arms: Placebo; REGN3500
Drug: Dupilumab — Administered SC q2w
  Other Names: REGN668; Dupixent
  Arms: Dupilumab; Placebo
Drug: REGN3500 + Dupilumab Combo — Administered SC q2w
  Other Names: REGN668; Dupixent
  Arms: Combo
Drug: Placebo — Administered SC q2w
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of REGN3500 monotherapy compared with placebo treatment in adult patients with moderate-to-severe Atopic dermatitis (AD).

Secondary Objectives are to:

* Evaluate the efficacy of REGN3500 in combination with dupilumab compared with placebo treatment in adult patients with moderate-to-severe AD
* Assess the safety, tolerability, and immunogenicity of subcutaneous (SC) doses of REGN3500 monotherapy and REGN3500 in combination with dupilumab in adult patients with moderate-to-severe AD
* Evaluate the Pharmacokinetic (PK) of REGN3500 monotherapy and REGN3500 in combination with dupilumab in adult patients with moderate-to-severe AD

ELIGIBILITY:
Key Inclusion Criteria:

1. Chronic AD, according to American Academy of Dermatology Consensus Criteria (Eichenfield, 2014), that has been present for at least 3 years before the screening visit
2. Eczema Area and Severity Index (EASI) score ≥16 at the screening and baseline visits
3. ≥10% Body surface area (BSA) of AD involvement at the screening and baseline visits
4. Documented recent history (within 6 months before the screening visit) of inadequate response to topical AD medication(s) or for whom topical treatments are medically inadvisable

Key Exclusion Criteria:

1. Prior participation in an anti-Interleukin (IL)-33 class antibody (including but not limited to REGN3500) or anti-IL-4Rα class antibody (including but not limited to dupilumab) clinical study; past treatment with or current treatment with dupilumab or another anti-IL-4Rα treatment
2. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit
3. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, tuberculosis (TB), histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per investigator judgment
4. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening
5. Positive with hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus antibody (HCV Ab) at the screening visit
6. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Note: Other protocol defined Inclusion/Exclusion Criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (51):
- United States (20):
  - Regeneron Research Site, Phoenix, Arizona
  - Regeneron Research Site, Fountain Valley, California
  - Regeneron Research Site, Long Beach, California
  - Regeneron Research Site, Los Angeles, California
  - Regeneron Research Site, Sacramento, California
  - Regeneron Research Site, Davie, Florida
  - Regeneron Research Site, Sandy Springs, Georgia
  - Regeneron Research Site, Rockville, Maryland
  - Regeneron Research Site, Bay City, Michigan
  - Regeneron Research Site, Saint Joseph, Michigan
  - Regeneron Research Site, Troy, Michigan
  - Regeneron Research Site, Forest Hills, New York
  - Regeneron Research Site, New York, New York
  - Regeneron Research Site, The Bronx, New York
  - Regeneron Research Site, High Point, North Carolina
  - Regeneron Research Site, Norman, Oklahoma
  - Regeneron Research Site, Portland, Oregon
  - Regeneron Research Site, Pittsburgh, Pennsylvania
  - Regeneron Research Site, Arlington, Texas
  - Regeneron Research Site, Richmond, Virginia
- Belgium (5):
  - Regeneron Research Site, Anderlecht
  - Regeneron Research Site, Antwerp
  - Regeneron Research Site, Brussels
  - Regeneron Research Site, Liège
  - Regeneron Research Site, Loverval
- Czechia (3):
  - Regeneron Research Site, Brno
  - Regeneron Research Site, Pardubice
  - Regeneron Research Site, Prague
- Germany (13):
  - Regeneron Research Site, Bad Bentheim
  - Regeneron Research Site, Berlin
  - Regeneron Research Site, Halle
  - Regeneron Research Site, Hamburg
  - Regeneron Research Site, Hanau
  - Regeneron Research Site, Leipzig
  - Regeneron Research Site, Lübeck
  - Regeneron Research Site, Mahlow
  - Regeneron Research Site, München
  - Regeneron Research Site, Münster
  - Regeneron Research Site, Quedlinburg
  - Regeneron Research Site, Tübingen
  - Regeneron Research Site, Witten
- Poland (5):
  - Regeneron Research Site, Bydgoszcz
  - Regeneron Research Site, Iwonicz-Zdrój
  - Regeneron Research Site, Krakow
  - Regeneron Research Site, Lodz
  - Regeneron Research Site, Wroclaw
- South Korea (3):
  - Regeneron Research Site, Gyeonggi-do
  - Regeneron Research Site, Incheon
  - Regeneron Research Site, Seoul
- Spain (2):
  - Regeneron Research Site, Barakaldo
  - Regeneron Research Site, Santiago de Compostela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 299 participants were screened at sites in Republic of Korea, United States of America, Germany, Poland, Czech Republic, Belgium and Spain. Out of 299 participants, 206 participants met eligibility criteria and randomized in this study.
Pre-assignment Details: Participants were randomized in a 1:1:1:1 ratio to 1 of the 4 treatment groups: Placebo every 2 weeks (Q2W); REGN3500 300 milligrams (mg) Q2W; Dupilumab 300 mg Q2W and combination of REGN3500 300 mg and Dupilumab 300 mg Q2W.
Groups:
- Placebo Q2W: Participants received 2 subcutaneous (SC) injections of placebo matched to REGN3500 and 2 SC injections of placebo matched to Dupilumab (loading dose) on Day 1 and then 2 SC injections of placebo matched to REGN3500 and 1 SC injection of placebo matched to Dupilumab Q2W up to Week 14.
- REGN3500 300 mg Q2W: Participants received 2 SC injections of REGN3500 at a dose of 150 mg (300 mg loading dose) and 2 SC injections of placebo matched to Dupilumab (loading dose) on Day 1 and then 2 SC injections of REGN3500 at a dose of 150 mg (300 mg loading dose) and 1 SC injection of placebo matched to Dupilumab Q2W up to Week 14.
- Dupilumab 300 mg Q2W: Participants received 2 SC injections of Dupilumab at a dose of 300 mg (600 mg loading dose) and 2 SC injections of placebo matched to REGN3500 on Day 1 and then 1 SC injection of Dupilumab at a dose 300 mg and 2 SC injections of placebo matched to REGN3500 Q2W up to Week 14.
- REGN3500 300 mg + Dupilumab 300 mg Q2W: Participants received 2 SC injections of REGN3500 at a dose of 150 mg (300 mg loading dose) and 2 SC injections of Dupilumab at a dose of 300 mg (600 mg loading dose) on Day 1 and then 2 SC injections of REGN3500 at a dose of 150 mg and 1 SC injection of Dupilumab at a dose of 300 mg Q2W up to Week 14.
Period: Overall Study
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Started | 51 | 52 | 51 | 52
Treated | 50 | 52 | 51 | 52
Completed | 20 | 24 | 27 | 22
Not Completed | 31 | 28 | 24 | 30
Not completed — Withdrawal by Subject | 26 | 25 | 23 | 26
Not completed — Lost to Follow-up | 3 | 2 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Randomized but never treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W | Total
Number analyzed (Participants) | 51 | 52 | 51 | 52 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (14.04) | 33.3 (12.19) | 38.4 (15.89) | 32.1 (12.10) | 34.7 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 23 | 22 | 80
  Male | 32 | 36 | 28 | 30 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 51 | 48 | 50 | 50 | 199
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 26 | 29 | 38 | 31 | 124
  Black or African American | 1 | 6 | 3 | 2 | 12
  Asian | 24 | 16 | 10 | 19 | 69
  Other | 0 | 1 | 0 | 0 | 1
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Scores on a Scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Population: FAS includes all randomized participants and was based on the treatment allocated (as randomized). Here, "Number of Participants Analyzed" signifies those participants who were evaluable at baseline.
  Scores on a Scale
    number analyzed (Participants) | 50 | 52 | 51 | 52 | 205
    (all) | 28.2 (9.54) | 29.9 (13.02) | 30.6 (13.86) | 29.0 (10.74) | 29.4 (11.87)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percent change from baseline in EASI score at Week 16 based on observed values set to missing after rescue treatment was reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: FAS included all randomized participants and was based on the treatment allocated (as randomized). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
  Due to premature discontinuation, all statistical analyses were descriptive, and no hypothesis testing was performed.
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 19 | 14 | 22 | 20
Percentage of Change | -52.4 (31.86) | -66.6 (22.46) | -77.8 (23.73) | -76.9 (20.79)

2. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percent change from baseline in EASI score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 23 | 23 | 26 | 24
Percentage of Change | -46.6 (36.58) | -58.0 (29.69) | -77.4 (22.59) | -75.8 (19.66)

3. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-50 (EASI-50) (Greater Than or Equal to [≥] 50 Percent [%] Improvement From Baseline) Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-50 (≥50% Improvement from baseline) at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 19 | 14 | 22 | 20
Percentage of Participants | 57.9 | 78.6 | 95.5 | 85.0

4. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-50 (EASI-50) (≥50% Improvement From Baseline) Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-50 (≥50% Improvement from baseline) at Week 16 were based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 23 | 23 | 26 | 24
Percentage of Participants | 52.2 | 65.2 | 96.2 | 87.5

5. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-75 (≥75% Improvement from baseline) at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders. Percentage of participants who achieved EASI-75 (>= 75% Improvement from baseline) at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 19 | 14 | 22 | 20
Percentage of Participants | 31.6 | 35.7 | 63.6 | 60.0

6. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-75 (≥75% Improvement from baseline) at Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 23 | 23 | 26 | 24
Percentage of Participants | 26.1 | 30.4 | 61.5 | 58.3

7. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-90 (EASI-90) (≥90% Improvement From Baseline) Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-90 (≥90% Improvement from baseline) at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 19 | 14 | 22 | 20
Percentage of Participants | 10.5 | 28.6 | 40.9 | 35.0

8. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-90 (EASI-90) (≥90% Improvement From Baseline) Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-90 (≥90% Improvement from baseline) at Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 23 | 23 | 26 | 24
Percentage of Participants | 8.7 | 17.4 | 38.5 | 29.2

9. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Absolute change from baseline in EASI score at Week 16 was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 19 | 14 | 22 | 20
Scores on a Scale | -13.25 (8.073) | -18.94 (9.383) | -25.40 (15.769) | -23.28 (9.177)

10. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Absolute change from baseline in EASI score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 23 | 23 | 26 | 24
Scores on a Scale | -12.18 (9.819) | -16.46 (10.002) | -24.06 (14.825) | -21.82 (9.008)

11. Secondary Outcome: Percentage of Participants With Both Investigator Global Assessment (IGA) Score 0 or 1 (on the 0 to 5 IGA Scale) and a Reduction From Baseline of ≥2 Points Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5 point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Participants with both IGA score of "0" or "1" and a reduction from baseline of >= 2 points at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing IGA score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 19 | 14 | 22 | 20
Percentage of Participants | 21.1 | 28.6 | 36.4 | 35.0

12. Secondary Outcome: Percentage of Participants With Both IGA Score 0 or 1 (on the 0 to 5 IGA Scale) and a Reduction From Baseline of ≥2 Points Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5 point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Participants with both IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 23 | 23 | 26 | 24
Percentage of Participants | 17.4 | 21.7 | 38.5 | 29.2

13. Secondary Outcome: Absolute Change From Baseline in Weekly Average of Daily Peak Pruritus Numerical Rating Scale (NRS) Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Absolute change from baseline in weekly average of daily Peak Pruritus NRS score at Week 16 based on observed values set to missing after rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 15 | 12 | 17 | 14
Scores on a Scale | -2.08 (2.825) | -2.90 (1.781) | -3.16 (2.607) | -3.92 (2.433)

14. Secondary Outcome: Absolute Change From Baseline in Weekly Average of Daily Peak Pruritus NRS Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Absolute change from baseline in weekly average of daily Peak Pruritus NRS score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 18 | 15 | 18 | 17
Scores on a Scale | -2.11 (2.651) | -2.87 (1.743) | -3.19 (2.532) | -3.64 (2.326)

15. Secondary Outcome: Percent Change From Baseline in in Weekly Average of Daily Peak Pruritus NRS Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percent change from baseline in weekly average of daily peak pruritus NRS score at Week 16 based on observed values set to missing after rescue treatment was reported. Values after first rescue treatment were set to missing and participants with missing NRS score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 15 | 12 | 17 | 14
Percentage of Change | -26.6 (36.71) | -38.0 (22.94) | -44.9 (35.73) | -60.2 (34.87)

16. Secondary Outcome: Percent Change From Baseline in in Weekly Average of Daily Peak Pruritus NRS Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percent change from baseline in weekly average of daily peak pruritus NRS score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 18 | 15 | 18 | 17
Percentage of Change | -27.6 (35.04) | -37.8 (21.88) | -45.1 (34.68) | -55.7 (34.22)

17. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) in Weekly Average of Peak Daily Pruritus NRS ≥4 Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percentage of participants with improvement of weekly average of daily peak pruritus NRS from baseline to Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing NRS at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 15 | 12 | 17 | 14
Percentage of Participants | 26.7 | 16.7 | 35.3 | 50.0

18. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) in Weekly Average of Peak Daily Pruritus NRS ≥4 Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percentage of participants with improvement of weekly average of daily peak pruritus NRS from baseline to Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 18 | 15 | 18 | 17
Percentage of Participants | 27.8 | 20.0 | 33.3 | 41.2

19. Secondary Outcome: Time to Onset of Effect on Pruritus (≥4-point Reduction of Weekly Average of Daily Peak Pruritus NRS From Baseline)
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?"
  Due to study discontinuation, not all planned participants were enrolled. For those already enrolled, the study drug was discontinued and participants were transitioned to post-treatment follow-up period. A large amount of data remained uncollected as not all enrolled participants completed all planned study visits and procedures for assessments for some endpoints. Therefore, this endpoint was removed and no data was collected for this outcome measure.
Time Frame: Week 16
Population: Due to premature discontinuation, all statistical analyses were descriptive, and no hypothesis testing was performed.
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) at Week 16
Description: The SCORAD index is a clinical tool for assessing the severity of atopic dermatitis (AD). Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
  Due to study discontinuation, not all planned participants were enrolled. For those already enrolled, the study drug was discontinued and participants were transitioned to post-treatment follow-up period. A large amount of data remained uncollected as not all enrolled participants completed all planned study visits and procedures for assessments for some endpoints. Therefore, this endpoint was removed and no data was collected for this outcome measure.
Time Frame: Week 16
Population: Due to premature discontinuation, all statistical analyses were descriptive, and no hypothesis testing was performed.
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Absolute Change From Baseline in Percent Body Surface Area (BSA) of Atopic Dermatitis (AD) Involvement at Week 16
Description: BSA affected by AD will be assessed for each section of the body using the rule of nines (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined. The proportion assigned to different body regions is different in younger children as compared to older children (head and neck area is assigned a higher proportion in younger children as compared to older children).
  Due to study discontinuation, not all planned participants were enrolled. For those already enrolled, the study drug was discontinued and participants were transitioned to post-treatment follow-up period. A large amount of data remained uncollected as not all enrolled participants completed all planned study visits and procedures for assessments for some endpoints. Therefore, this endpoint was removed and no data was collected for this outcome measure.
Time Frame: Week 16
Population: Due to premature discontinuation, all statistical analyses were descriptive, and no hypothesis testing was performed.
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs) From Baseline up to Week 16
Description: Adverse Event (AE): any untoward medical occurrence in a participant administered a study drug which may/may not have a causal relationship with study drug. Serious AE (SAE): any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAE: AEs starting/worsening after first intake of study drug. TEAEs included: SAEs and Non-SAEs. AESI included: Anaphylactic reactions; Systemic/severe hypersensitivity reactions; Malignancy; Helminthic infections; Suicide-related events; Severe injection site reactions; Mycosis fungoides/other forms of cutaneous T-cell lymphoma; any clinical endoparasitosis; Conjunctivitis and significant Alanine aminotransferase (ALT) elevation. Number of participants with TEAEs, Serious TEAES and AESIs from baseline up to Week 16 were reported.
Time Frame: Baseline up to Week 16
Population: Safety analysis set (SAF) included all randomized participants who received any study drug and was based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 50 | 52 | 51 | 52
Participants
  Participants with TEAEs | 25 | 24 | 29 | 22
  Participants with Serious TEAEs | 1 | 0 | 1 | 1
  Participants with AESIs | 2 | 0 | 1 | 2

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs) From Baseline up to Week 36
Description: AE: any untoward medical occurrence in a participant administered a study drug which may/may not have a causal relationship with study drug. SAE: any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAE: AEs starting/worsening after first intake of study drug. TEAEs included both SAEs and Non-SAEs. AESI included: Anaphylactic reactions; Systemic/severe hypersensitivity reactions; Malignancy; Helminthic infections; Suicide-related events; Severe injection site reactions; Mycosis fungoides/other forms of cutaneous T-cell lymphoma; any clinical endoparasitosis; Conjunctivitis and significant ALT elevation. Number of participants with TEAEs, Serious TEAES and AESIs from baseline up to Week 36 were reported.
Time Frame: Baseline up to Week 36
Population: SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 50 | 52 | 51 | 52
Participants
  Participants with TEAEs | 27 | 26 | 35 | 28
  Participants with Serious TEAEs | 1 | 1 | 2 | 1
  Participants with AESIs | 2 | 0 | 1 | 2

24. Secondary Outcome: Number of Participants With Positive Treatment-Emergent Anti-drug Antibodies (ADA) to REGN3500 and Dupilumab
Description: Treatment-Emergent (TE) ADA: any positive post baseline assay response when baseline results were negative/missing. TE ADA responses were further classified as: - persistent (treatment-emergent positive ADA response detected in at least 2 consecutive post baseline samples separated by at least a 16-week post baseline period [based on nominal sampling time], with no ADA-negative samples in-between, regardless of any missing samples or a positive response at the last ADA sampling time point),- indeterminate (a positive assay response at the last collection time point only, regardless of any missing samples), - transient (not persistent/indeterminate, regardless of any missing samples). Here, "Number of Participants Analysed" signifies those participants who were evaluable for this endpoint.
Time Frame: Baseline up to Week 36
Population: The ADA analysis set (AAS) included all participants who received any study drug and had at least 1 non-missing ADA result in the respective ADA assays, after the first dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | REGN3500 300 mg Q2W | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 43 | 48 | 44 | 46
Participants | 0 | 0 | 3 | 6

25. Secondary Outcome: Serum Concentration of Functional REGN3500
Description: Serum Concentration of Functional REGN3500 was reported. Data was reported for REGN3500 300 mg Q2W and REGN3500 300 mg + Dupilumab 300 mg Q2W arms only
Time Frame: Baseline (Week 0), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, and 36
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received any study drug (active or placebo [safety analysis set]) and who had at least 1 non-missing study drug concentration result following the first dose of study drug. Here, "Number Analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | REGN3500 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 52 | 52
Milligrams per Liter (mg/L)
  Week 0 | 0 (0) | 0.00373 (0.0269)
  Week 2: number analyzed (Participants) | 52 | 51
  Week 2 | 22.8 (9.06) | 25.2 (9.58)
  Week 4: number analyzed (Participants) | 48 | 46
  Week 4 | 41.6 (14.8) | 41.9 (16.4)
  Week 8: number analyzed (Participants) | 39 | 43
  Week 8 | 58.8 (20.5) | 63.0 (22.8)
  Week 12: number analyzed (Participants) | 30 | 36
  Week 12 | 67.4 (26.7) | 74.5 (25.7)
  Week 16: number analyzed (Participants) | 16 | 21
  Week 16 | 73.9 (31.4) | 82.4 (33.5)
  Week 20: number analyzed (Participants) | 9 | 15
  Week 20 | 33.3 (21.9) | 45.1 (24.2)
  Week 24: number analyzed (Participants) | 8 | 11
  Week 24 | 13.1 (11.9) | 23.3 (14.4)
  Week 28: number analyzed (Participants) | 5 | 11
  Week 28 | 7.31 (5.49) | 12.3 (12.5)
  Week 32: number analyzed (Participants) | 6 | 10
  Week 32 | 4.61 (4.48) | 5.43 (4.12)
  Week 36: number analyzed (Participants) | 7 | 11
  Week 36 | 2.42 (2.70) | 2.79 (2.48)

26. Secondary Outcome: Serum Concentration of Functional Dupilumab
Description: Serum Concentration of Functional Dupilumab was reported.
Time Frame: Baseline (Week 0), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, and 36
Population: Data were reported for Dupilumab 300 gm Q2W and REGN3500 300 mg + Dupilumab 200 mg Q2W arms only. Pharmacokinetic (PK) analysis set included all randomized participants who received any study drug (active or placebo [safety analysis set]) and who had at least 1 non-missing study drug concentration result following the first dose of study drug. Here, "Number Analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dupilumab 300 mg Q2W | REGN3500 300 mg + Dupilumab 300 mg Q2W
Number analyzed (Participants) | 51 | 52
mg/L
  Week 0 | 0 (0) | 0.00219 (0.0158)
  Week 2: number analyzed (Participants) | 50 | 51
  Week 2 | 51.4 (19.0) | 50.6 (19.0)
  Week 4: number analyzed (Participants) | 47 | 46
  Week 4 | 51.5 (23.6) | 57.6 (26.1)
  Week 8: number analyzed (Participants) | 40 | 43
  Week 8 | 63.0 (32.5) | 64.9 (26.3)
  Week 12: number analyzed (Participants) | 37 | 36
  Week 12 | 70.4 (37.8) | 69.6 (29.2)
  Week 16: number analyzed (Participants) | 23 | 21
  Week 16 | 73.4 (39.2) | 71.6 (30.9)
  Week 20: number analyzed (Participants) | 15 | 15
  Week 20 | 25.8 (26.9) | 28.0 (24.8)
  Week 24: number analyzed (Participants) | 14 | 11
  Week 24 | 4.36 (8.97) | 6.50 (12.5)
  Week 28: number analyzed (Participants) | 14 | 11
  Week 28 | 1.47 (3.86) | 2.39 (7.93)
  Week 32: number analyzed (Participants) | 14 | 10
  Week 32 | 0.0227 (0.0850) | 0 (0)
  Week 36: number analyzed (Participants) | 11 | 11
  Week 36 | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the end of study (Week 36) regardless of seriousness or relationship to investigational product (IP).
Groups:
- R3500 300 mg Q2W: Participants received 2 SC injections of REGN3500 at a dose of 150 mg (300 mg loading dose) and 2 SC injections of placebo matched to Dupilumab (loading dose) on Day 1 and then 2 SC injections of REGN3500 at a dose of 150 mg (300 mg loading dose) and 1 SC injection of placebo matched to Dupilumab Q2W up to Week 14.
- R3500 300 mg and Dupilumab 300 mg Q2W: Participants received 2 SC injections of REGN3500 at a dose of 150 mg (300 mg loading dose) and 2 SC injections of Dupilumab at a dose of 300 mg (600 mg loading dose) on Day 1 and then 2 SC injections of REGN3500 at a dose of 150 mg and 1 SC injection of Dupilumab at a dose of 300 mg Q2W up to Week 14.
Arm/Group | Placebo Q2W | R3500 300 mg Q2W | Dupilumab 300 mg Q2W | R3500 300 mg and Dupilumab 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52 | 0/51 | 1/52
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/52 | 2/51 | 1/52
Other Adverse Events (participants affected / at risk) | 17/50 | 15/52 | 25/51 | 20/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (N=50) | R3500 300 mg Q2W (N=52) | Dupilumab 300 mg Q2W (N=51) | R3500 300 mg and Dupilumab 300 mg Q2W (N=52)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goodpasture's syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (N=50) | R3500 300 mg Q2W (N=52) | Dupilumab 300 mg Q2W (N=51) | R3500 300 mg and Dupilumab 300 mg Q2W (N=52)
Nasopharyngitis (Infections and infestations) | 8 (9) | 5 (5) | 11 (14) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 3 (4)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (9) | 7 (8) | 8 (11) | 10 (11)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The decision was made by the sponsor to terminate the study on 12 Feb 2020 due to lack of efficacy. Study enrollment was not complete at that time, therefore planned sample sizes were not met. Participants discontinued study drug and transitioned into the post-treatment follow-up period. As a result of the decision to terminate the study, all statistical analyses were descriptive and no hypothesis testing was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03736967/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03736967/SAP_001.pdf